CLINICAL TRIAL: NCT05181176
Title: Effect of Coffee and Tea Consumption on Adolescent Weight Control - a Randomized Clinical Trial
Brief Title: Effect of Coffee and Tea Consumption on Adolescent Weight Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TLV-18-0166
Record Dates: First submitted 2021-12-06; First posted 2022-01-06 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2021-12

CONDITIONS: Body Weight
Keywords: Obesity
MeSH Terms: conditions — Body Weight; Obesity | interventions — Coffee; Tea; Teas, Herbal

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, parallel group study comparing 3 weight loss interventions comprised of a similar dietary recommendation with either coffee (coffee group), tea (tea group) or placebo (herbal tea).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coffee (Experimental): The coffee group was instructed to consume 2 cups of coffee a day, the amount that was previously described as beneficial in epidemiological studies and safe for children and adolescence. Each cup of coffee contains 250 ml of coffee, which contains approximately 80 mg of caffeine. The children were allowed to add milk to the coffee and sweeten it with artificial sweetener
  Interventions: Dietary Supplement: Coffee
- Green Tea (Experimental): The green tea group will be instructed to drink 3 cups (230CC) of Chinese green tea (Wissotzky Tea Israel Ltd). Each tea bag contains 500 g of fine dried herb parts. Each cup contains 84 mg total catechin and 32 mg caffeine. The participants were instructed to leave the tea bag for 2 minutes before drinking.
  Interventions: Dietary Supplement: Green tea
- Herbal tea (Placebo Comparator): The control group consumed 3 cups a day of Wissotzky- kid drink (Wissotzky Tea Israel Ltd), which is a drink that is marketed for children containing an infusion of fruits and plants. Each tea bag contains 2.7 gr plants parts with no evidence of polyphenols or caffeine.
  Interventions: Dietary Supplement: Herbal tea (placebo)

INTERVENTIONS:
Dietary Supplement: Coffee — 3 weight-loss interventions comprised of a similar dietary recommendation with either coffee (coffee group), tea (tea group) or placebo (herbal tea).
  Arms: Coffee
Dietary Supplement: Green tea — 3 weight-loss interventions comprised of a similar dietary recommendation with either coffee (coffee group), tea (tea group) or placebo (herbal tea).
  Arms: Green Tea
Dietary Supplement: Herbal tea (placebo) — 3 weight-loss interventions comprised of a similar dietary recommendation with either coffee (coffee group), tea (tea group) or placebo (herbal tea).
  Arms: Herbal tea

SUMMARY:
Introduction: The influence of tea or coffee supplementation on body weight in adolescents has never been tested. The aim of the present study was to investigate the effect of tea and coffee consumption on body weight and body fat in an obese adolescent population.

Methods: Randomized clinical trial, parallel group study comparing 3 weight loss interventions comprised of a similar dietary recommendation with either coffee (coffee group), tea (tea group) or placebo (herbal tea). Sociodemographic data and medical history details were retrieved from medical files. The body mass index Z (BMI Z) score and fat percentage as measured by bioelectrical impedance were compared between groups at 3 and 6 months.

DETAILED DESCRIPTION:
Patient Population The participants were recruited at the at the Obesity Clinic in the Pediatric Gastroenterology Unit at "Dana Dwek" Children's Hospital from January 2018 and December 2020. The Obesity Clinic is a tertiary referral center for children and adolescent with obesity and its complication. Adolescents aged 12-17 years with BMI in the 95th percentile or higher were eligible for the study. Exclusion criteria included major medical, chronic use of medication that may affect study outcomes or regular intake of some tea or coffee (individual for whom the intervention would likely produce relatively little change in habitual intake).

Study Design This is a randomized clinical trial, parallel-group study comparing 3 weight loss interventions comprising standardized dietary recommendation either with coffee (coffee group) tea (tea group) or placebo (herbal tea). The study consists of 2 weeks run in period and 24 weeks treatment period.

Intervention The 3 groups received similar weight reducing interventions comprising diets that will differentiated only with regard to the recommendation for coffee or green tea consumption. The standard intervention included 2 weekly family-based counseling concerning nutritional education (low carbohydrate, low glycemic index diet), behavioral counseling and physical activity.

The coffee group instructed to consume 2 cups of coffee a day, amount that was previously describe as beneficial in epidemiological studies and safe for children and adolescence. Each cup of coffee contains 250 ml of coffee, which contains approximately 80 mg of caffeine. The children were allowed to add milk to the coffee and sweeten it with artificial sweetener.

The green tea group will be instructed to drink 3 cups (230CC) of Chinese green tea (Wissotzky Tea Israel Ltd). Each tea bag contains 500 g fine dried herb parts. Each cup contains 84 mg total catechin and 32 mg caffeine. The participants were instructed to leave the tea bag for 2 minutes before drinking. The control group consumed 3 cups a day of Wissotzky- kid drink (Wissotzky Tea Israel Ltd), which is a drink that is marketed for children containing infusion of fruits and plants. Each tea bag contains 2.7 gr plants parts with no evidence of polyphenols or caffeine.

The tea was provided to the participants and adherence was ensured by 3 days dietary questioners at each visit and by collecting empty boxes every month.

Outcomes

Information retrieved from medical files of subjects included:

1. Sociodemographic characteristics: age, sex
2. Medical history: perinatal characteristics (birth weight, gestational age), medications and family history of cardio-metabolic diseases (diabetes, hypertension, dyslipidemia, cardiovascular disease, and cerebrovascular episodes) in first- and second-degree relatives.
3. Physical examination: systolic and diastolic BP and anthropometric measurements (height, weight, calculated BMI and body fat)
4. Screening for obesity-related comorbidities: laboratory metabolic workup, abdominal ultrasonography (steatohepatitis) and polysomnography findings (obstructive sleep apnea).

The primary outcomes of the study were decrease in BMI Z score, Percentile and body fat at 3 and 6 months of the intervention.

Weight and height was assessed at baseline and monthly for 3-month period and again after 6 month. Body weight and fat percentage was indirectly measured by BIA (Tanita Body-Composition Analyzer, Tanita DC-360 S and GMON Professional Software), which has been clinically verified to be accurate and reliable and to provide highly reproducible results. The GMON software provides the BIA data adjusted for sex, age, height, and race (Caucasian and Asian) according to reference ranges 12The BMI Z score and percentile was calculated using reference data for sex and age. Metabolic parameters documented upon admission included glucose, insulin, HDL, LDL, TG, ALT AST CRP. Fatty liver and fibrosis was assessed by ultrasonography. At each monthly visit the participant provided 3-day dietary questionnaire.

Definition of Study Variables BMI percentiles and Z-scores of anthropometric measurements were calculated with PediTools Electronic Growth Chart Calculators based upon CDC growth charts. The height, weight, and BMI values were converted to sex- and age-specific z-scores according to the CDC 2000 growth charts. Weight status was defined according to the BMI z-score as follows: overweight as a BMI percentile ≥85th and <95th percentiles (1.036 ≤BMI z-score <1.645), and obese as a BMI percentile ≥95th percentile (BMI z-score ≥1.645).

Childhood MetS components were defined as follows: glucose intolerance = fasting glucose ≥100 mg/dL (5.5 mmol/L); elevated BP = systolic and/or diastolic BP ≥90th percentile for sex, age, and height; hypertriglyceridemia = triglyceride (TG) levels ≥110 mg/dL (1.24 mmol/L), and low high-density lipoprotein-cholesterol (HDL-c) = HDL-c ≤40 mg/dL (1.03 mmol/L).

Obesity-related comorbidities were compiled as follows. Insulin resistance was the calculation of Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) by fasting insulin μU/mL x fasting glucose mmol/L/22.5. The healthy range for HOMA-IR was defined as a value between 0.5-1.4, early insulin resistance was defined as a value ≥1.9, and significant insulin resistance was defined as a value ≥2.9. Nonalcoholic fatty liver disease (NAFLD) was suspected in a child with typical clinical features (obesity and persistent mild elevations of serum alanine aminotransferase [ALT] >2 x upper limit of normal). A provisional diagnosis of NAFLD was made by excluding other causes of liver disease through a focused history, physical examination, laboratory evaluation, and an abdominal ultrasound showing increased echogenicity suggestive of fatty liver. Obstructive sleep apnea was defined by recurrent events of partial or complete upper airway obstruction during sleep as detected by polysomnography performed in patients with a history of persistent snoring and/or recurrent awakenings. Pseudotumor cerebri was diagnosed according to the modified Dandy criteria: symptoms and signs of increased intracranial pressure (e.g., headache, transient visual obscurations, papilledema, visual loss), no other neurologic abnormalities, elevated intracranial pressure with normal cerebrospinal fluid composition, and a neuroimaging study that shows no etiology for intracranial hypertension .

Statistical Analyses SPSS (IBM Corp. Released 2016. IBM SPSS Statistics for Windows, Version 27.0. Armonk, NY: IBM Corp.) was used for all statistical analysis.

All statistical tests were two-sided. The Kolmogorov-Smirnov test and the Shapiro-Wilk test were applied to assess the normality of continuous data. The data are expressed as means±SDs for normally distributed variables and median and interquartile range [IQR] for skewed distribution. Pearson's chi-square test was performed to compare the distribution of categorical variables between 3 intervention group. Kruskal wallis test followed by Dunn's post hoc test was used to compare the differences between Coffee Tea and placebo for continuous variable . The changes over time were compared for each arm separately using Friedman's test for paired data followed by Dunn's post hoc test. A P value ≤0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-17 years with BMI in the 95th percentile or higher were eligible for the study.

Exclusion Criteria:

* Exclusion criteria included major medical, chronic use of medication that may affect study outcomes or regular intake of some tea or coffee (individual for whom the intervention would likely produce relatively little change in habitual intake).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
effect tea and coffee consumption on body weight | 6 months
  change in BMI Z score

SECONDARY OUTCOMES:
effect tea and coffee consumption on body fat | 6 months
  change in fat percentage analysis using bio electrical impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hadar Moran Lev, MD, Principal Investigator — Pediatric Gastroenterology
Locations (1):
- Pediatric Gastroenterology Unit, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
the individual participant data will be anonymous to other researchers

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Tobias DK, Chen M, Manson JE, Ludwig DS, Willett W, Hu FB. Effect of low-fat diet interventions versus other diet interventions on long-term weight change in adults: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2015 Dec;3(12):968-79. doi: 10.1016/S2213-8587(15)00367-8. Epub 2015 Oct 30. PMID 26527511
- [Background] Wadden TA, Stunkard AJ, Liebschutz J. Three-year follow-up of the treatment of obesity by very low calorie diet, behavior therapy, and their combination. J Consult Clin Psychol. 1988 Dec;56(6):925-8. doi: 10.1037//0022-006x.56.6.925. No abstract available. PMID 3204204
- [Background] Kramer FM, Jeffery RW, Forster JL, Snell MK. Long-term follow-up of behavioral treatment for obesity: patterns of weight regain among men and women. Int J Obes. 1989;13(2):123-36. PMID 2663745
- [Background] Pasman WJ, Westerterp-Plantenga MS, Muls E, Vansant G, van Ree J, Saris WH. The effectiveness of long-term fibre supplementation on weight maintenance in weight-reduced women. Int J Obes Relat Metab Disord. 1997 Jul;21(7):548-55. doi: 10.1038/sj.ijo.0800439. PMID 9226484
- [Background] Mukhtar H, Ahmad N. Tea polyphenols: prevention of cancer and optimizing health. Am J Clin Nutr. 2000 Jun;71(6 Suppl):1698S-702S; discussion 1703S-4S. doi: 10.1093/ajcn/71.6.1698S. PMID 10837321
- [Background] Khan N, Mukhtar H. Tea polyphenols for health promotion. Life Sci. 2007 Jul 26;81(7):519-33. doi: 10.1016/j.lfs.2007.06.011. Epub 2007 Jun 28. PMID 17655876
- [Background] Butt MS, Sultan MT. Green tea: nature's defense against malignancies. Crit Rev Food Sci Nutr. 2009 May;49(5):463-73. doi: 10.1080/10408390802145310. PMID 19399671
- [Background] Nagao T, Hase T, Tokimitsu I. A green tea extract high in catechins reduces body fat and cardiovascular risks in humans. Obesity (Silver Spring). 2007 Jun;15(6):1473-83. doi: 10.1038/oby.2007.176. PMID 17557985
- [Background] Murase T, Nagasawa A, Suzuki J, Hase T, Tokimitsu I. Beneficial effects of tea catechins on diet-induced obesity: stimulation of lipid catabolism in the liver. Int J Obes Relat Metab Disord. 2002 Nov;26(11):1459-64. doi: 10.1038/sj.ijo.0802141. PMID 12439647
- [Background] Zheng G, Sayama K, Okubo T, Juneja LR, Oguni I. Anti-obesity effects of three major components of green tea, catechins, caffeine and theanine, in mice. In Vivo. 2004 Jan-Feb;18(1):55-62. PMID 15011752
- [Background] Lin JK, Lin-Shiau SY. Mechanisms of hypolipidemic and anti-obesity effects of tea and tea polyphenols. Mol Nutr Food Res. 2006 Feb;50(2):211-7. doi: 10.1002/mnfr.200500138. PMID 16404708
- [Background] Auvichayapat P, Prapochanung M, Tunkamnerdthai O, Sripanidkulchai BO, Auvichayapat N, Thinkhamrop B, Kunhasura S, Wongpratoom S, Sinawat S, Hongprapas P. Effectiveness of green tea on weight reduction in obese Thais: A randomized, controlled trial. Physiol Behav. 2008 Feb 27;93(3):486-91. doi: 10.1016/j.physbeh.2007.10.009. Epub 2007 Oct 18. PMID 18006026
- [Background] Westerterp-Plantenga MS, Lejeune MP, Kovacs EM. Body weight loss and weight maintenance in relation to habitual caffeine intake and green tea supplementation. Obes Res. 2005 Jul;13(7):1195-204. doi: 10.1038/oby.2005.142. PMID 16076989
- [Background] Hursel R, Westerterp-Plantenga MS. Green tea catechin plus caffeine supplementation to a high-protein diet has no additional effect on body weight maintenance after weight loss. Am J Clin Nutr. 2009 Mar;89(3):822-30. doi: 10.3945/ajcn.2008.27043. Epub 2009 Jan 28. PMID 19176733
- [Background] Wan CJ, Lin LY, Yu TH, Sheu WH. Metabolic syndrome associated with habitual indulgence and dietary behavior in middle-aged health-care professionals. J Diabetes Investig. 2010 Dec 3;1(6):259-65. doi: 10.1111/j.2040-1124.2010.00055.x. PMID 24843441
- [Background] Higdon JV, Frei B. Coffee and health: a review of recent human research. Crit Rev Food Sci Nutr. 2006;46(2):101-23. doi: 10.1080/10408390500400009. PMID 16507475
- [Background] Wu T, Willett WC, Hankinson SE, Giovannucci E. Caffeinated coffee, decaffeinated coffee, and caffeine in relation to plasma C-peptide levels, a marker of insulin secretion, in U.S. women. Diabetes Care. 2005 Jun;28(6):1390-6. doi: 10.2337/diacare.28.6.1390. PMID 15920057
- [Background] Odegaard AO, Pereira MA, Koh WP, Arakawa K, Lee HP, Yu MC. Coffee, tea, and incident type 2 diabetes: the Singapore Chinese Health Study. Am J Clin Nutr. 2008 Oct;88(4):979-85. doi: 10.1093/ajcn/88.4.979. PMID 18842784
- [Background] Greenberg JA, Axen KV, Schnoll R, Boozer CN. Coffee, tea and diabetes: the role of weight loss and caffeine. Int J Obes (Lond). 2005 Sep;29(9):1121-9. doi: 10.1038/sj.ijo.0802999. PMID 15925959
- [Background] Lopez-Garcia E, van Dam RM, Rajpathak S, Willett WC, Manson JE, Hu FB. Changes in caffeine intake and long-term weight change in men and women. Am J Clin Nutr. 2006 Mar;83(3):674-80. doi: 10.1093/ajcn.83.3.674. PMID 16522916
- [Background] Brener A, Peleg I, Rosenfeld T, Kern S, Uretzky A, Elkon-Tamir E, Rosen G, Levinson H, Israeli G, Interator H, Lebenthal Y. Beyond Body Mass Index - Body Composition Assessment by Bioimpedance in Routine Endocrine Practice. Endocr Pract. 2021 May;27(5):419-425. doi: 10.1016/j.eprac.2020.10.013. Epub 2020 Dec 15. PMID 33934752
- [Background] Shypailo RJ, Motil KJ. The Use of Bioimpedance in Pediatric Health, Nutrition, and Disease. J Pediatr Gastroenterol Nutr. 2018 Oct;67(4):435-436. doi: 10.1097/MPG.0000000000002068. No abstract available. PMID 30239486
- [Background] Kuczmarski RJ, Ogden CL, Guo SS, Grummer-Strawn LM, Flegal KM, Mei Z, Wei R, Curtin LR, Roche AF, Johnson CL. 2000 CDC Growth Charts for the United States: methods and development. Vital Health Stat 11. 2002 May;(246):1-190. PMID 12043359
- [Background] Ogden CL, Flegal KM. Changes in terminology for childhood overweight and obesity. Natl Health Stat Report. 2010 Jun 25;(25):1-5. PMID 20939253
- [Background] Flynn JT, Kaelber DC, Baker-Smith CM, Blowey D, Carroll AE, Daniels SR, de Ferranti SD, Dionne JM, Falkner B, Flinn SK, Gidding SS, Goodwin C, Leu MG, Powers ME, Rea C, Samuels J, Simasek M, Thaker VV, Urbina EM; SUBCOMMITTEE ON SCREENING AND MANAGEMENT OF HIGH BLOOD PRESSURE IN CHILDREN. Clinical Practice Guideline for Screening and Management of High Blood Pressure in Children and Adolescents. Pediatrics. 2017 Sep;140(3):e20171904. doi: 10.1542/peds.2017-1904. Epub 2017 Aug 21. PMID 28827377
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S13-S28. doi: 10.2337/dc19-S002. PMID 30559228
- [Background] Vos MB, Abrams SH, Barlow SE, Caprio S, Daniels SR, Kohli R, Mouzaki M, Sathya P, Schwimmer JB, Sundaram SS, Xanthakos SA. NASPGHAN Clinical Practice Guideline for the Diagnosis and Treatment of Nonalcoholic Fatty Liver Disease in Children: Recommendations from the Expert Committee on NAFLD (ECON) and the North American Society of Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN). J Pediatr Gastroenterol Nutr. 2017 Feb;64(2):319-334. doi: 10.1097/MPG.0000000000001482. PMID 28107283
- [Background] Bitners AC, Arens R. Evaluation and Management of Children with Obstructive Sleep Apnea Syndrome. Lung. 2020 Apr;198(2):257-270. doi: 10.1007/s00408-020-00342-5. Epub 2020 Mar 12. PMID 32166426
- [Background] Vardi P, Shahaf-Alkalai K, Sprecher E, et al. Components of the metabolic syndrome (MTS), hyperinsulinemia, and insulin resistance in obese Israeli children and adolescents. Diabetes Metab Syndr Clin Res Rev. 2007;1(2):97-103
- [Derived] Moran-Lev H, Cohen S, Zelber-Sagi S, Mazkeret Mayer E, Anafy A, Yerushalmy-Feler A, Lubetzky R. Effect of Coffee and Tea Consumption on Adolescent Weight Control: An Interventional Pilot Study. Child Obes. 2023 Mar;19(2):121-129. doi: 10.1089/chi.2022.0032. Epub 2022 May 30. PMID 35639365